CLINICAL TRIAL: NCT00064064
Title: A Phase II Study of Triapine in Combination With Gemcitabine in Patients With Metastatic Non-Small Cell Lung Cancer
Brief Title: 3-AP and Gemcitabine in Treating Patients With Metastatic Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vion Pharmaceuticals (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000306462; VION-CLI-030; MDA-ID-030143
Record Dates: First submitted 2003-07-08; First posted 2003-07-09 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2004-08

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Gemcitabine; 3-aminopyridine-2-carboxaldehyde thiosemicarbazone

INTERVENTIONS:
Drug: gemcitabine hydrochloride
Drug: triapine

SUMMARY:
RATIONALE: Drugs used in chemotherapy such as gemcitabine use different ways to stop tumor cells from dividing so they stop growing or die. 3-AP may stop the growth of tumor cells by blocking the enzymes necessary for tumor cell growth and may help gemcitabine kill more cancer cells by making them more sensitive to the drug.

PURPOSE: Phase II trial to study the effectiveness of combining gemcitabine with 3-AP in treating patients who have metastatic non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the partial and complete objective response rate in patients with metastatic non-small cell lung cancer treated with 3-AP and gemcitabine.
* Determine the progression-free and overall survival in patients treated with this regimen.
* Determine the safety of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive 3-AP IV over 4 hours followed by gemcitabine IV over 30 minutes once weekly on weeks 1-3. Treatment repeats every 4 weeks for up to 12 courses in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 22-50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer

  * Metastatic disease
* Progressive disease after no more than 2 prior cytotoxic regimens containing at least 1 of the following drugs:

  * Cisplatin
  * Carboplatin
  * Taxane
  * Vinorelbine
* Measurable disease
* No CNS metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Life expectancy

* More than 3 months

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 9 g/dL (transfusion allowed)

Hepatic

* Bilirubin no greater than 2.0 mg/dL
* ALT and AST no greater than 3 times upper limit of normal (ULN) (5 times ULN if liver metastases present)
* Chronic viral hepatitis allowed

Renal

* Creatinine no greater than 2.0 mg/dL

Cardiovascular

* No myocardial infarction within the past 3 months
* No uncontrolled congestive heart failure
* No uncontrolled coronary artery disease
* No uncontrolled cardiac arrhythmias

Pulmonary

* No dyspnea at rest
* No supplemental oxygen dependence

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study participation
* No active infection
* No other prior or concurrent malignancy except carcinoma in situ of the cervix previously treated by cone biopsy and/or resection, nonmetastatic basal cell or squamous cell skin cancer, or any stage I malignancy curatively resected more than 5 years ago
* No other concurrent life-threatening illness

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Prior non-cytotoxic biologic regimens allowed (e.g., vaccines, antibodies, cytokines, or small molecule cell signaling inhibitors)

Chemotherapy

* See Disease Characteristics
* More than 3 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* No prior gemcitabine
* No prior 3-AP

Endocrine therapy

* Not specified

Radiotherapy

* More than 4 weeks since prior radiotherapy and recovered

Surgery

* More than 3 weeks since prior surgery and recovered

Other

* More than 3 weeks since prior non-cytotoxic regimens

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-01; Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mario Sznol, MD, Study Chair — Vion Pharmaceuticals
Locations (5):
- United States (4):
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Sarah Cannon Cancer Center at Centennial Medical Center, Nashville, Tennessee
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
- University Medical Center Nijmegen, Nijmegen, Netherlands